CLINICAL TRIAL: NCT00768768
Title: A Study of Skin/Nail Sensation and the Pharmacokinetics of the Uptake of Terbinafine in the Great Toe Nail and Systemically Following Treatment With the Electrokinetic Transungual System (ETS)-Terbinafine Gel in Healthy Normal Voluneteers
Brief Title: Iontophoretic Application of Terbinafine Gel to the Large Toe Nail
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Transport Pharmaceuticals (Industry)
Responsible Party: Craig Sprenger, MD, Cetero Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPI-N-111
Record Dates: First submitted 2008-10-06; First posted 2008-10-08 (Estimated); Last update posted 2009-03-12 (Estimated); Status verified 2009-03

CONDITIONS: Onychomycosis
Keywords: iontophoresis; terbinafine; onychomycosis
MeSH Terms: conditions — Onychomycosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Active Comparator): Iontophoretic Dose Level 1
  Interventions: Other: Electrokinetic Transungual System (ETS) - Terbinafine Gel
- 2 (Active Comparator): Iontophoretic Dose Level 2
  Interventions: Other: ETS-Terbinafine Gel
- 3 (Active Comparator): Iontophoretic Dose Level 3
  Interventions: Other: ETS-Terbinafine Gel
- 4 (Active Comparator): Iontophoretic Dose Level 4
  Interventions: Other: ETS-Terbinafine Gel
- 5 (Active Comparator): Iontophoretic Dose Level 5
  Interventions: Other: ETS-Terbinafine Gel

INTERVENTIONS:
Other: Electrokinetic Transungual System (ETS) - Terbinafine Gel — Iontophoresis in conjunction with a terbinafine gel
  Drug Dose: ETS drug cartridge loaded with approximately 20 mg - 35 mg of terbinafine in the gel formulation, with the load depending on the size of the toenail to be treated.
  Two different drug applicators to be tested on each subject
  Single treatment on each toenail; one treatment with one drug applicator design, the second treatment with the alternative drug applicator design
  Iontophoretic Dose: 3 mA-min as 0.3 mA for 10 min
  Arms: 1
Other: ETS-Terbinafine Gel — Iontophoresis in conjunction with a terbinafine gel
  Drug Dose: ETS drug cartridge loaded with approximately 20 mg - 35 mg of terbinafine in the gel formulation, with the load depending on the size of the toenail to be treated.
  Two different drug applicators to be tested on each subject
  Single treatment on each toenail; one treatment with one drug applicator design, the second treatment with the alternative drug applicator design
  Iontophoretic Dose: 6 mA-min as 0.5 mA for 12 min
  Arms: 2
Other: ETS-Terbinafine Gel — Iontophoresis in conjunction with a terbinafine gel
  Drug Dose: ETS drug cartridge loaded with approximately 20 mg - 35 mg of terbinafine in the gel formulation, with the load depending on the size of the toenail to be treated.
  Two different drug applicators to be tested on each subject
  Single treatment on each toenail; one treatment with one drug applicator design, the second treatment with the alternative drug applicator design
  Iontophoretic Dose: 6 mA-min as 0.3 mA for 20 min
  Arms: 3
Other: ETS-Terbinafine Gel — Iontophoresis in conjunction with a terbinafine gel
  Drug Dose: ETS drug cartridge loaded with approximately 20 mg - 35 mg of terbinafine in the gel formulation, with the load depending on the size of the toenail to be treated.
  Two different drug applicators to be tested on each subject
  Single treatment on each toenail; one treatment with one drug applicator design, the second treatment with the alternative drug applicator design
  Iontophoretic Dose: 10 mA-min as 0.5 mA for 20 min
  Arms: 4
Other: ETS-Terbinafine Gel — Iontophoresis in conjunction with a terbinafine gel
  Drug Dose: ETS drug cartridge loaded with approximately 20 mg - 35 mg of terbinafine in the gel formulation, with the load depending on the size of the toenail to be treated.
  Two different drug applicators to be tested on each subject
  Single treatment on each toenail; one treatment with one drug applicator design, the second treatment with the alternative drug applicator design
  Iontophoretic Dose: 15 mA-min as 0.5 mA for 30 min
  Arms: 5

SUMMARY:
Terbinafine is recognized as one of the most effective drugs for the treatment of toe nail fungus (onychomycosis). This trial will be the first test of a new device to improve the delivery of terbinafine directly to the toe nail. The device uses a low level of electric current, iontophoresis, to "push" the terbinafine into the nail.

The study will involve a single application of terbinafine, in a gel form, with the iontophoretic device. The treatment will be applied to the surface of both large toenails of healthy subjects. Subjects will be asked to report any sensations in the nail or surrounding skin experienced during or after treatment. Samples from the edge of the treated toe nail will be taken at 2-4 week intervals to measure how much terbinafine was delivered to the nails, and blood samples will be taken for the first 24 hours after treatment to determine how much, if any, terbinafine was absorbed into the subjects's body. Observations will also be made of the treated toes to look for any irritation of the surrounding skin due to the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers between 18 and 75 years of age, inclusive.

Exclusion Criteria:

* Subjects with pacemakers or automatic implantable cardioverter/defibrillator
* Subjects with an implantable electronic device.
* Subjects with a history of diabetes.
* Subjects with a history of onychomycosis or an abnormal appearing nail on the great toe
* Subject using systemic antifungal medications within 6 months prior to study enrollment.
* Subject using prescription topical antifungal medications for toenail fungus within 3 months or other commercially available medications for toenail fungus applied directly to the toenail within 1 week prior to study enrollment.
* Subject with a history of allergic or adverse response to terbinafine or any related anti-fungal drug
* Participation in a previous clinical trial involving an investigational drug or device within 30 days prior to study enrollment.
* Subject requires chronic use of analgesics, pain medication, or non-steroidal anti-inflammatory agents (NSAIDS).
* In females of childbearing potential, a positive urine pregnancy test at screening and just prior to dosing.
* Nursing mothers.
* Subject with a history of alcoholism or drug abuse within the preceding 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Evaluate the skin/nail sensation noted by subjects during and following iontophoretic application of terbinafine gel to the great toenail | 12 weeks

SECONDARY OUTCOMES:
Evaluate the uptake into the nail of the great toe and the systemic uptake and pharmacokinetics of terbinafine following a single iontophoretic application of terbinafine gel | 12 weeks and 24 hours, respectively

CONTACTS AND LOCATIONS:
Overall Officials: Craig Sprenger, MD, Principal Investigator — Cetero Research, San Antonio; Eric M Morrel, PhD, Study Director — Transport Pharmaceuticals, Inc.; Philip M Friden, PhD, Study Director — Transport Pharmaceuticals, Inc.
Locations (1):
- Cetero Research, Fargo, North Dakota, United States